CLINICAL TRIAL: NCT03916406
Title: A PHASE 1, RANDOMIZED, OPEN LABEL, 2-WAY CROSSOVER STUDY TO EVALUATE THE EFFECT OF REPEATED DOSING OF PF-06835919 ON THE PHARMACOKINETICS OF A SINGLE ORAL DOSE OF MIDAZOLAM IN HEALTHY PARTICIPANTS
Brief Title: THE EFFECT OF MULTIPLE DOSES OF PF-06835919 ON THE PHARMACOKINETICS OF A SINGLE ORAL MIDAZOLAM DOSE IN HEALTHY PARTICIPANTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C1061016; 2019-000929-42 (EudraCT Number)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): midazolam alone followed by combination of PF 06835919 and midazolam
  Interventions: Drug: PF 06835919; Drug: Midazolam
- Sequence 2 (Experimental): PF 06835919 in combination with midazolam followed by midazolam alone
  Interventions: Drug: PF 06835919; Drug: Midazolam

INTERVENTIONS:
Drug: PF 06835919 — 300 mg
Drug: Midazolam — 7.5 mg

SUMMARY:
This is a Phase 1, randomized, open label, 2 way crossover drug drug interaction (DDI) study which will evaluate the impact of PF 06835919 on midazolam pharmacokinetics in healthy participants. Participants will be randomized to 1 of 2 treatment sequences as described below. A total of approximately 10 healthy male and/or female participants will be enrolled in this study so that approximately 5 participants will be enrolled into each treatment sequence. In this crossover study, 2 treatments are being assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiovascular tests.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed
* Participants, who according to the product label for midazolam, would be at increased risk if dosed with midazolam (ie, including but not limited to participants with history of myasthenia gravis, chronic obstructive pulmonary disease (COPD), pulmonary insufficiency, glaucoma, concomitant central nervous system (CNS) depressants).
* History of hypersensitivity to midazolam or any other benzodiazepine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
AUCinf of midazolam following a single oral dose | Baseline up to 51 days
  Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf)

SECONDARY OUTCOMES:
AUClast of midazolam following a single oral dose. | Baseline up to 51 days
  Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Cmax of midazolam following a single oral dose. | Baseline up to 51 days
  Maximum Observed Plasma Concentration (Cmax)
Incidence of Adverse Events in participants | Screening up to 79 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Be-bru, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1061016&StudyName=A+PHASE+1%2C+RANDOMIZED%2C+OPEN+LABEL%2C+2-WAY+CROSSOVER+STUDY+TO+EVALUATE+THE+EFFECT+OF+REPEATED+DOSING+OF+PF-06835919+ON+THE+PHARMACOKINETICS+OF+A+SINGLE+ORAL+DOSE+OF+MIDAZOLAM+IN+HEALTHY+PARTICIPANTS